CLINICAL TRIAL: NCT04676724
Title: A Phase IIb Multi-Center, Randomised, Open Label Study to Assess the Efficacy and Safety of Sequential Treatment With GSK3228836 Followed by Pegylated Interferon Alpha 2a in Participants With Chronic Hepatitis B Virus (B-Together)
Brief Title: Study of Sequential GSK3228836 and Peginterferon Treatment in Participants With Chronic Hepatitis B (CHB)
Acronym: B-Together
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209348
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis B
Keywords: Chronic Hepatitis B; GSK3228836; Pegylated interferon; Nucleos(t)ide analogue; Sustained virologic response
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a ratio of 1:1 to one of two treatment arms: 24 weeks GSK3228836 followed by up to 24 weeks PegIFN, or 12 weeks GSK3228836 followed by up to 24 weeks PegIFN.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3228836 300 mg (24 weeks) + PegIFN 180 mcg (24 weeks) (Experimental): Participants on stable NA therapy received 300 milligrams per week (mg/week) GSK3228836 for 24 weeks (plus a loading dose on Day 4 and 11), followed by Pegylated Interferon (PegIFN) 180 microgram per week (mcg/week) up to 24 weeks.
  Interventions: Drug: GSK3228836; Drug: PegIFN; Drug: NA therapy
- GSK3228836 300 mg (12 weeks) + PegIFN 180 mcg (24 weeks) (Experimental): Participants on stable NA therapy received 300mg/week GSK3228836 for 12 weeks (plus a loading dose on Day 4 and 11), followed by PegIFN 180 mcg/week up to 24 weeks.
  Interventions: Drug: GSK3228836; Drug: PegIFN; Drug: NA therapy

INTERVENTIONS:
Drug: GSK3228836 — Participants will be administered GSK3228836.
Drug: PegIFN — Participants will be administered PegIFN.
Drug: NA therapy — Participants will continue to receive their NA therapy for the duration of the study.

SUMMARY:
This study is intended to evaluate if 12 or 24 weeks of treatment with GSK3228836 followed by up to 24 weeks of pegylated interferon (PegIFN) can increase the rate of hepatitis B virus surface antigen (HBsAg) loss in participants on stable nucleos(t)ide analogue (NA) therapy, and whether virologic response can be sustained once PegIFN treatment is discontinued. Participants will be randomized to receive GSK3228836 for 12 or 24 weeks followed by up to 24 weeks of PegIFN.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age at the time of signing the informed consent.
* Participants who are eligible to be treated with PegIFN.
* Documented chronic HBV infection >=6 months prior to screening and currently receiving stable NA therapy except telbivudine, defined as no changes to their NA regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study.
* Plasma or serum HBsAg concentration >100 International Units per milliliter (IU/mL).
* Plasma or serum HBV DNA concentration <90 IU/mL.
* ALT <=2 times ULN.
* A male participant is eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of study treatment: a) Refrain from donating sperm; b) Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or agree to use contraception/barrier: Agree to use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak) when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* A female participant is eligible to participate: a) If she is not pregnant or breastfeeding; b) at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1 percent per year), preferably with low user dependency during the intervention period and for at least 90 days after the last dose of study treatment.
* A WOCBP must have both a negative highly sensitive pregnancy test within 24 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative, a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Clinically significant abnormalities, aside from chronic HBV infection in medical history or physical examination.
* Co-infection with: Current or past history of Hepatitis C virus (HCV); Human immunodeficiency virus (HIV); Hepatitis D virus (HDV).
* History of or suspected liver cirrhosis and/or evidence of cirrhosis as determined by both: Aspartate aminotransferase (AST)-Platelet Index (APRI) >2 and FibroSure/FibroTest result >0.7. If only one parameter (APRI or FibroSure/FibroTest) result is positive, a discussion with the Medical Monitor is required before inclusion in study is permitted. Regardless of APRI of Fibrosure/FibroTest score, if the participant meets one of the following criteria, they will be excluded from the study: a) Liver biopsy (i.e., Metavir Score F4); b) Liver stiffness >12 kilopascals (kPa).
* Diagnosed or suspected hepatocellular carcinoma as evidenced by the following: Alpha- fetoprotein concentration >=200 nanogram per milliliter (ng/mL); If the screening alpha fetoprotein concentration is >=50 ng/mL and <200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before randomization.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer). Participants under evaluation for possible malignancy are not eligible.
* History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause) or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
* Poorly controlled thyroid dysfunction or abnormal thyroid stimulating hormone (TSH) levels
* Positive (or borderline positive) anti-neutrophil cytoplasmic antibody (ANCA) at screening. Participants that meet these criteria may be considered for inclusion in the study following: a) Analysis of myeloperoxidase (MPO)-ANCA [perinuclear ANCA (pANCA)] and PR3-ANCA [classical ANCA (cANCA)]; b) A discussion with the Medical Monitor to review participant's complete medical history to ensure no past history or current manifestations of a vasculitic/inflammatory/auto-immune condition.
* Low complement 3 (C3) at screening and evidence of past history or current manifestations of vasculitic/inflammatory/auto-immune conditions. All participants with low C3 at screening should have their medical history discussed with the Medical Monitor prior to enrolment.
* History of alcohol or drug abuse/dependence. Current alcohol use as judged by investigator to potentially interfere with participant compliance; History of or current drug abuse/dependence as judged by the investigator to potentially interfere with participant compliance. Refers to illicit drugs and substances with abuse potential. Medications that are used by the participant as directed, whether over-the-counter or through prescription, are acceptable and would not meet the exclusion criteria.
* Pre-existing severe psychiatric condition or a history of severe psychiatric disorders, including severe depression, suicidal ideation and attempted suicide.
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
* Participants for whom immunosuppressive treatment is not advised, including therapeutic doses of steroids, will be excluded.
* Participants with prior treatment with PegINF or interferon will be excluded
* Participants requiring anti-coagulation therapies (for example warfarin, Factor Xa inhibitors or anti-platelet agents like clopidogrel).
* Participants currently taking, or took within 6 months of screening, telbivudine.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives (if known) or twice the duration (if known) of the biological effect of the study treatment (whichever is longer) or 90 days (if half-life or duration is unknown).
* Prior treatment with any oligonucleotide or small interfering ribonucleic acid (siRNA) within 12 months prior to the first dosing day.
* Fridericia's QT correction formula (QTcF) >=450 milliseconds (msec) (if single electrocardiogram [ECG] at screening shows QTcF>=450 msec, a mean of triplicate measurements should be used to confirm that participant meets exclusion criterion).
* Laboratory results as follows: Serum albumin <3.5 grams per deciliter (g/dL); Glomerular filtration rate (GFR) <60 milliliter per minute per 1.73 square meter (mL/min /1.73 m^2) as calculated by the Chronic Kidney Disease Epidemiologic Collaboration (CKD-EPI) formula (for Japan, Japanese Society of Nephrology Chronic Kidney Disease Initiative [JSN-CKDI equation]); International normalized ratio (INR) >1.25; Platelet count <140x10^9 cells/L; Baseline hemoglobin <10 g/dL; Total bilirubin >1.25 times ULN (For participants with benign unconjugated hyperbilirubinemia with total bilirubin >1.25 times ULN, discussion for inclusion to the study is required with the Medical Monitor); Urine albumin to creatinine ratio (ACR) >=0.03 milligram (mg)/mg (or >=30 mg/g). In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement. In cases where participants have low urine albumin and low urine creatinine levels resulting in a urine ACR calculation >=0.03 mg/mg (or >=30 mg/g), the investigator should confirm that the participant does not have a history of diabetes, hypertension or other risk factors that may affect renal function and discuss with the Medical Monitor, or designee.
* History of/sensitivity to GSK3228836 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (45):
- United States (4):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New York, New York
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Montreal, Quebec
- China (4):
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
- Italy (3):
  - GSK Investigational Site, Baggiovara (MO), Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza (MB), Lombardy
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Tokyo
- Poland (3):
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Łańcut
- Russia (7):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Красноярск
- South Africa (2):
  - GSK Investigational Site, Ennerdale, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Ulsan
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santander
- United Kingdom (4):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Joshi S, Freudenberg JM, Singh JM, Jordan WT, Felton L, Dixon S, Paff M, Theodore D, Walker J. Immunomodulation by bepirovirsen may induce killing of infected hepatocytes (B-Together study). Hepatol Int. 2025 Oct 3. doi: 10.1007/s12072-025-10917-0. Online ahead of print. PMID 41042426
- [Derived] Buti M, Heo J, Tanaka Y, Andreone P, Atsukawa M, Cabezas J, Chak E, Coffin CS, Fujiwara K, Gankina N, Gordon SC, Janczewska E, Komori A, Lampertico P, McPherson S, Morozov V, Plesniak R, Poulin S, Ryan P, Sagalova O, Sheng G, Voloshina N, Xie Q, Yim HJ, Dixon S, Paff M, Felton L, Lee M, Greene T, Lim J, Lakshminarayanan D, McGonagle G, Plein H, Youssef AS, Elston R, Kendrick S, Theodore D. Sequential Peg-IFN after bepirovirsen may reduce post-treatment relapse in chronic hepatitis B. J Hepatol. 2025 Feb;82(2):222-234. doi: 10.1016/j.jhep.2024.08.010. Epub 2024 Aug 29. PMID 39214467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 108 participants were enrolled in this study.
Pre-assignment Details: Participants who were on stable nucleos(t)ide analogue (NA) therapy randomized (1:1) into one of 2 parallel treatment arms. Treatment arm 1: 300 mg/week GSK3228836 for 24 weeks + PegIFN 180 mcg/week for 24 weeks; on-treatment until Week 48 and off-treatment from Weeks 48 to 72. Treatment arm 2: 300 mg/week GSK3228836 for 12 weeks + 180 mcg/week PegIFN for 24 weeks, on-treatment until Week 36 and off-treatment follow-up from Weeks 36 to Week 60 and 72.
Period: Overall Study
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Started | 55 | 53
Completed | 49 | 50
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks): Participants on stable NA therapy received 300mg/week GSK3228836 for 24 weeks (plus a loading dose on Day 4 and 11), followed by PegIFN 180 microgram per week (mcg/week) up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks) | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 45.5 (10.73) | 45.5 (9.35) | 45.5 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 44 | 33 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 30 | 26 | 56
  BLACK OR AFRICAN AMERICAN | 3 | 3 | 6
  WHITE | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Treatment Arm 1 - Percentage of Participants Achieving Sustained Virologic Response (SVR) for 24 Weeks After End of Treatment
Description: Sustained virologic response is defined as undetectable levels of Hepatitis B surface antigen (HBsAg) and Hepatitis-B virus deoxy-ribonucleic acid (HBV DNA) on treatment. The SVR was a composite endpoint defined as HBsAg and HBV DNA levels were less than (<) Lower limit of quantitation (LLOQ) at the planned end of sequential treatment of GSK3228836 and PegIFN treatment which is sustained for 24 weeks post-GSK3228836 and PegIFN treatment in the absence of any rescue medication. Percentage values are rounded-off.
Time Frame: Up to 24 weeks off treatment (Study Weeks 48 to 72)
Population: Intent to Treat (ITT) Set that included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
Percentage of Participants | 9

2. Primary Outcome: Treatment Arm 2 - Percentage of Participants Achieving Sustained Virologic Response (SVR) for 24 Weeks After End of Treatment
Description: as for outcome 1
Time Frame: Up to 24 weeks off treatment (Study Weeks 36 to 60)
Population: Intent to Treat (ITT) Set that included all randomized participants. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Percentage of Participants | 15

3. Secondary Outcome: Treatment Arm 1: Percentage of Participants Achieving HBsAg and HBV DNA < Lower Limit of Quantitation (LLOQ)
Description: Percentage of participants achieving HBsAg and HBV DNA <LLOQ were reported. Percentage values are rounded-off.
Time Frame: End of treatment (up to 48 weeks) and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Percentage of Participants
  End of treatment (up to 48 weeks): number analyzed (Participants) | 38
  End of treatment (up to 48 weeks) | 15
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 13

4. Secondary Outcome: Treatment Arm 2: Percentage of Participants Achieving HBsAg and HBV DNA < Lower Limit of Quantitation (LLOQ)
Description: Percentage of participants achieving HBsAg and HBV DNA <LLOQ were reported. Percentage values are rounded-off.
Time Frame: End of treatment (up to 36 weeks), up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) and up to 36 weeks off treatment follow-up (Study Weeks 36 to 72)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 50
Percentage of Participants
  End of treatment (up to 36 weeks): number analyzed (Participants) | 36
  End of treatment (up to 36 weeks) | 15
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 17
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 15

5. Secondary Outcome: Treatment Arm 1: Percentage of Participants With Categorical Changes From Baseline in HBsAg Values
Description: Participants who achieved a decline in HBsAg values from baseline were reported. Participants were categorized in the following categorical HBsAg decline of <0.5, greater than or equal to (>=) 0.5, >=1, >=1.5, and >=3 log10 international units per milliliter (IU/mL). The 'HBsAg < LLOQ' category is derived based on Absolute/raw HBsAg result. The HBsAg decline categories are based on change from baseline values. Percentage values are rounded-off.
Time Frame: Baseline, End of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Percentage of Participants
  HBsAg <LLOQ - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg <LLOQ - End of Treatment (up to 48 weeks) | 18
  HBsAg<LLOQ - Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 13
  HBsAg decline <0.5 - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg decline <0.5 - End of Treatment (up to 48 weeks) | 24
  HBsAg decline <0.5- Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 45
  HBsAg decline >=0.5 - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg decline >=0.5 - End of Treatment (up to 48 weeks) | 42
  HBsAg decline >=0.5 - Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 44
  HBsAg decline >=1 - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg decline >=1 - End of Treatment (up to 48 weeks) | 33
  HBsAg decline >=1- Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 36
  HBsAg decline >=1.5 - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg decline >=1.5 - End of Treatment (up to 48 weeks) | 27
  HBsAg decline >=1.5 - Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 36
  HBsAg decline >=3 - End of Treatment (up to 48 weeks): number analyzed (Participants) | 38
  HBsAg decline >=3 - End of Treatment (up to 48 weeks) | 20
  HBsAg decline >=3 - Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 27

6. Secondary Outcome: Treatment Arm 2: Percentage of Participants With Categorical Changes From Baseline in HBsAg Values
Description: as for outcome 5
Time Frame: Baseline, End of treatment (up to 36 weeks), up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) and up to 36 weeks off treatment follow-up (Study Weeks 36 to 72)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 50
Percentage of Participants
  HBsAg <LLOQ - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg <LLOQ - End of Treatment (up to 36 weeks) | 15
  HBsAg<LLOQ - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 17
  HBsAg <LLOQ - Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 15
  HBsAg decline <0.5 - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg decline <0.5 - End of Treatment (up to 36 weeks) | 26
  HBsAg decline <0.5 - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 42
  HBsAg decline <0.5 - Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 43
  HBsAg decline >=0.5 - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg decline >=0.5 - End of Treatment (up to 36 weeks) | 42
  HBsAg decline >=0.5 - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 51
  HBsAg decline >=0.5 - Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 47
  HBsAg decline >=1 - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg decline >=1 - End of Treatment (up to 36 weeks) | 34
  HBsAg decline >=1 - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 34
  HBsAg decline >=1 - Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 32
  HBsAg decline >=1.5 - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg decline >=1.5 - End of Treatment (up to 36 weeks) | 28
  HBsAg decline >=1.5 - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 23
  HBsAg decline >=1.5-up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 19
  HBsAg decline >=3 - End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  HBsAg decline >=3 - End of Treatment (up to 36 weeks) | 15
  HBsAg decline >=3 - Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 17
  HBsAg decline >=3 - Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 17

7. Secondary Outcome: Treatment Arm 1: Number of Participants With Alanine Aminotransferase (ALT) Normalization
Description: The ALT normalization (ALT <=upper limit of normal [ULN]) over time in absence of rescue medication in participants with baseline ALT>ULN and ALT data at that visit. Participants who achieved ALT normalization were reported.
Time Frame: At baseline, end of treatment (up to 48 weeks) and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: Intent to Treat (ITT) Set that included all randomized participants. The "n" represents the number of participants with baseline ALT > ULN and ALT data at that visit. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
Participants
  ALT>ULN, At Baseline | 4
  ALT normalization, End of Treatment (up to 48 weeks): number analyzed (Participants) | 4
  ALT normalization, End of Treatment (up to 48 weeks) | 0
  ALT normalization, Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 4
  ALT normalization, Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 2

8. Secondary Outcome: Treatment Arm 2: Number of Participants With Alanine Aminotransferase (ALT) Normalization
Description: as for outcome 7
Time Frame: At baseline, End of treatment (up to 36 weeks), up to 24 weeks off treatment follow-up (Study Weeks 36 to 60), and up to 36 weeks off treatment follow-up (Study Weeks 36 to 72)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Participants
  ALT>ULN, At Baseline | 10
  ALT normalization, End of Treatment (up to 36 weeks): number analyzed (Participants) | 7
  ALT normalization, End of Treatment (up to 36 weeks) | 1
  ALT normalization, Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 9
  ALT normalization, Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 5
  ALT normalization, Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 9
  ALT normalization, Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 6

9. Secondary Outcome: Treatment Arm 1: Number of Participants With HBe Antibody (Anti-HBeAg) Levels
Description: Blood samples were collected to assess HBe antibody levels and results reported are for baseline HBeAg positive participants.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 13
Participants
  At Baseline | 2
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 9
  End of Treatment (up to 48 weeks) | 5
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 4

10. Secondary Outcome: Treatment Arm 2: Number of Participants With HBe Antibody (Anti-HBeAg) Levels
Description: as for outcome 9
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 14
Participants
  At Baseline | 1
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 9
  End of Treatment (up to 36 weeks) | 1
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 1
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 0

11. Secondary Outcome: Treatment Arm 1: Mean Change From Baseline in HBe Antibody Levels
Description: Blood samples were collected to assess HBe antibody levels and results reported are for baseline HBeAg positive participants. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 14
Log10 IU/mL
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 9
  End of Treatment (up to 48 weeks) | -1.04 (1.133)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 13
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | -0.81 (1.044)

12. Secondary Outcome: Treatment Arm 2: Mean Change From Baseline in HBe Antibody Levels
Description: as for outcome 11
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 13
Log10 IU/mL
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 9
  End of Treatment (up to 36 weeks) | -0.52 (0.598)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 12
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | -0.58 (0.766)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | -0.65 (0.787)

13. Secondary Outcome: Treatment Arm 1: Actual Values of HBsAg Levels
Description: Blood samples were collected from participants to assess HBsAg at indicated time points.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
Log10 IU/mL
  At Baseline | 3.34 (0.555)
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 48 weeks) | 1.52 (2.071)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 1.72 (2.043)

14. Secondary Outcome: Treatment Arm 2: Actual Values of HBsAg Levels
Description: Blood samples were collected from participants to assess HBsAg at indicated time points.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Log10 IU/mL
  At Baseline | 3.32 (0.622)
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 36 weeks) | 1.70 (1.896)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 2.12 (1.827)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 2.12 (1.830)

15. Secondary Outcome: Treatment Arm 1: Mean Change From Baseline in HBsAg Levels
Description: Blood samples were collected to assess HBsAg change from baselines levels. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Log10 IU/mL
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 48 weeks) | -1.76 (1.726)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | -1.58 (1.722)

16. Secondary Outcome: Treatment Arm 2: Mean Change From Baseline in HBsAg Levels
Description: as for outcome 15
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Log10 IU/mL
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 36 weeks) | -1.54 (1.567)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | -1.20 (1.458)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | -1.20 (1.460)

17. Secondary Outcome: Treatment Arm 1: Actual Values of HBV DNA Levels
Description: Blood samples were collected to assess HBV DNA levels.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
Log10 IU/mL
  At Baseline | 0.64 (0.796)
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 35
  End of Treatment (up to 48 weeks) | 0.97 (0.629)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 47
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 0.17 (0.438)

18. Secondary Outcome: Treatment Arm 2: Actual Values of HBV DNA Levels
Description: Blood samples were collected to assess HBV DNA levels.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Log10 IU/mL
  At Baseline | 0.57 (0.687)
  End of treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of treatment (up to 36 weeks) | 0.70 (0.700)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 0.34 (0.579)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 0.35 (0.587)

19. Secondary Outcome: Treatment Arm 1: Mean Change From Baseline in HBV DNA Levels
Description: Blood samples were collected to assess HBV DNA levels. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 47
Log10 IU/mL
  End of treatment (up to 48 weeks): number analyzed (Participants) | 35
  End of treatment (up to 48 weeks) | 0.40 (0.945)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | -0.39 (0.727)

20. Secondary Outcome: Treatment Arm 2: Mean Change From Baseline in HBV DNA Levels
Description: as for outcome 19
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Log10 IU/mL
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of Treatment (up to 36 weeks) | 0.21 (0.925)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | -0.21 (0.876)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | -0.22 (0.754)

21. Secondary Outcome: Treatment Arm 1: Actual Values of Hepatitis B Virus E-antigen (HBeAg) Levels
Description: Blood samples were collected to assess HBeAg levels.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
Log10 IU/mL
  At Baseline | 14.221 (69.3438)
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 10
  End of Treatment (up to 48 weeks) | 0.250 (0.4193)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 15
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 1.197 (2.4945)

22. Secondary Outcome: Treatment Arm 2: Actual Values of Hepatitis B Virus E-antigen (HBeAg) Levels
Description: Blood samples were collected to assess HBeAg levels.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Log10 IU/mL
  At Baseline | 8.510 (42.1588)
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 12
  End of Treatment (up to 36 weeks) | 3.008 (6.2682)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 14
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 3.410 (6.0421)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 15
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 2.797 (4.8973)

23. Secondary Outcome: Treatment Arm 1: Mean Change From Baseline in HBeAg Levels
Description: Blood samples were collected to assess HBeAg levels. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 15
Log10 IU/mL
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 10
  End of Treatment (up to 48 weeks) | -21.774 (65.4276)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | -19.482 (55.1948)

24. Secondary Outcome: Treatment Arm 2: Mean Change From Baseline in HBeAg Levels
Description: as for outcome 23
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 15
Log10 IU/mL
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 12
  End of Treatment (up to 36 weeks) | -5.270 (8.8942)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 14
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | -26.384 (80.2108)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | -26.345 (77.2836)

25. Secondary Outcome: Treatment Arm 1: Actual Values of HBs Antibody Levels
Description: Blood samples were collected to assess HBs antibody levels.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/L
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 54
Log10 IU/L
  At Baseline | 0.62 (0.271)
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 48 weeks) | 1.06 (0.903)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 0.82 (0.718)

26. Secondary Outcome: Treatment Arm 2: Actual Values of HBs Antibody Levels
Description: Blood samples were collected to assess HBs antibody levels.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/L
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
Log10 IU/L
  At Baseline | 0.69 (0.204)
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of Treatment (up to 36 weeks) | 0.87 (0.491)
  Up to 24 weeks off treatment follow-up (study week 36 to week 60): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (study week 36 to week 60) | 0.80 (0.521)
  Up to 36 weeks off treatment follow-up (study week 36 to week 72): number analyzed (Participants) | 49
  Up to 36 weeks off treatment follow-up (study week 36 to week 72) | 0.76 (0.481)

27. Secondary Outcome: Treatment Arm 1: Mean Change From Baseline in HBs Antibody Levels
Description: Blood samples were collected to assess HBs antibody levels over time. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/L
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 48
Log10 IU/L
  End of treatment (up to 48 weeks): number analyzed (Participants) | 35
  End of treatment (up to 48 weeks) | 0.42 (0.934)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 0.18 (0.757)

28. Secondary Outcome: Treatment Arm 2: Mean Change From Baseline in HBs Antibody Levels
Description: as for outcome 27
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 IU/L
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
Log10 IU/L
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of Treatment (up to 36 weeks) | 0.18 (0.450)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 0.09 (0.487)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 0.05 (0.453)

29. Secondary Outcome: Treatment Arm 1: Actual Values of ALT
Description: Blood samples were collected to assess ALT mean values.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International Units Per Liter (IU/L)
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55
International Units Per Liter (IU/L)
  At Baseline | 22.7 (13.97)
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 48 weeks) | 53.1 (60.61)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | 19.2 (9.77)

30. Secondary Outcome: Treatment Arm 2: Actual Values of ALT
Description: Blood samples were collected to assess ALT mean values.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 53
IU/L
  At Baseline | 26.9 (19.16)
  End of Treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of Treatment (up to 36 weeks) | 55.3 (46.60)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60): number analyzed (Participants) | 49
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | 22.1 (13.30)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | 23.5 (15.61)

31. Secondary Outcome: Treatment Arm 1: Change From Baseline in ALT
Description: Blood samples were collected to assess ALT values. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At baseline, end of treatment (up to 48 weeks), and up to 24 weeks off treatment follow-up (Study Weeks 48 to 72)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
IU/L
  End of Treatment (up to 48 weeks): number analyzed (Participants) | 36
  End of Treatment (up to 48 weeks) | 27.6 (56.05)
  Up to 24 weeks off treatment follow-up (Study Weeks 48 to 72) | -3.8 (9.86)

32. Secondary Outcome: Treatment Arm 2: Change From Baseline in ALT
Description: as for outcome 31
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 49
IU/L
  End of treatment (up to 36 weeks): number analyzed (Participants) | 35
  End of treatment (up to 36 weeks) | 27.8 (40.55)
  Up to 24 weeks off treatment follow-up (Study Weeks 36 to 60) | -4.3 (17.50)
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72): number analyzed (Participants) | 48
  Up to 36 weeks off treatment follow-up (Study Weeks 36 to 72) | -3.1 (18.65)

33. Secondary Outcome: Treatment Arm 1 - Median Time to ALT Normalization in Absence of Rescue Medication for 24 Weeks After End of Treatment
Description: Time to ALT normalization in absence of rescue medication were measured in participants having Baseline ALT>ULN.
Time Frame: Up to 24 weeks off treatment (Study Week 48 to72)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 4
Weeks | NA [6.3 to NA] — The estimate for Median Time to Event (Weeks) is not estimable (NE) for Arm 1 because the survival curve did not reach below 0.5 at the last timepoint. The corresponding 95% CI's upper limit is NE because the number of events in Arm 1 was too small to provide an estimate.

34. Secondary Outcome: Treatment Arm 2 - Median Time to ALT Normalization in Absence of Rescue Medication for 24 Weeks After End of Treatment
Description: Time to ALT normalization in absence of rescue medication were measured in participants having Baseline ALT>ULN.
Time Frame: Up to 24 weeks off treatment (Study Weeks 36 to 60)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 10
Weeks | 4.1 [1.1 to 47.1]

35. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response (SVR) for 24 Weeks Off Treatment for Comparison of Efficacy Between Different Treatment Durations
Description: Sustained virologic response is defined as undetectable levels of HBsAg and Hepatitis-B virus deoxy-ribonucleic acid (HBV DNA) on treatment. The SVR was a composite endpoint defined as Hepatitis B surface antigen (HBsAg) and Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) levels were less than (<) Lower limit of quantitation (LLOQ) at the planned end of GSK3228836 treatment which is sustained for 24 weeks post-GSK3228836 treatment in the absence of rescue medication. The point estimate for the difference in SVR and its respective credible interval (CI) were evaluated at 24 weeks off of planned treatment for both arms. The comparison of efficacy is between treatment durations and timepoint corresponds to Week 72 in Arm 1 and Week 60 in Arm 2. 95% CI here refers as credible interval. Percentage values are rounded-off.
Time Frame: Up to 24 weeks off treatment (Treatment Arm 1: Study Weeks 48 to 72 and Treatment Arm 2: Study Weeks 36 to 60)
Population: Intent to Treat (ITT) Set that included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
Number analyzed (Participants) | 55 | 53
Percentage of participants | 9 | 15
Statistical Analysis 1: Comparison: GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) vs GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks); Test type: Other; Difference in SVR Rate = -3, 95% CI 2-sided [-29 to 11] — The point estimate of SVR and its 95% highest posterior density Credible Interval (CI) are estimated from a Bayesian model that incorporates the analysis stratification factors and treatment arm

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: All-cause mortality, Serious adverse events and non-serious adverse events were reported for the Safety Population who were randomized and received at least one dose of study treatment.
Arm/Group | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 6/55 | 2/53
Other Adverse Events (participants affected / at risk) | 52/55 | 50/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) (N=55) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks) (N=53)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3228836 300 mg (24 Weeks) + PegIFN 180 mcg (24 Weeks) (N=55) | GSK3228836 300 mg (12 Weeks) + PegIFN 180 mcg (24 Weeks) (N=53)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 10 (18) | 7 (10)
Neutropenia (Blood and lymphatic system disorders) | 10 (25) | 12 (21)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (20) | 11 (16)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (12) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (8) | 4 (4)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (14) | 6 (6)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Asthenia (General disorders) | 5 (8) | 10 (21)
Chills (General disorders) | 3 (5) | 1 (2)
Discomfort (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (19) | 5 (8)
Influenza like illness (General disorders) | 12 (14) | 8 (12)
Malaise (General disorders) | 7 (11) | 3 (3)
Pain (General disorders) | 2 (7) | 2 (2)
Pyrexia (General disorders) | 17 (25) | 14 (19)
Vaccination site pain (General disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (5) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 15 (15) | 5 (5)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (2)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (3)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (7)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 4 (5)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 2 (6)
Alanine aminotransferase increased (Investigations) | 23 (36) | 6 (9)
Antineutrophil cytoplasmic antibody increased (Investigations) | 1 (1) | 1 (2)
Antineutrophil cytoplasmic antibody positive (Investigations) | 1 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 16 (21) | 6 (6)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 3 (3) | 4 (8)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Complement factor C3 decreased (Investigations) | 7 (9) | 3 (3)
Complement factor C4 decreased (Investigations) | 8 (11) | 2 (2)
Complement fragment Bb increased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 6 (35) | 4 (24)
Creatinine renal clearance increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 1 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2)
Hepatitis B DNA increased (Investigations) | 2 (2) | 0 (0)
Monocyte chemotactic protein-1 increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 14 (22) | 8 (12)
Platelet count decreased (Investigations) | 10 (13) | 5 (5)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Thyroxine increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 2 (5)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 8 (14) | 4 (7)
Cell death (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (9) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 12 (25)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4)
Headache (Nervous system disorders) | 7 (29) | 12 (25)
Hypoaesthesia (Nervous system disorders) | 1 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Muscle contractions involuntary (Nervous system disorders) | 2 (2) | 1 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (8)
Tremor (Nervous system disorders) | 1 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Hyposomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (6)
Irritability (Psychiatric disorders) | 1 (1) | 3 (4)
Libido decreased (Psychiatric disorders) | 1 (1) | 2 (2)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (5)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Injection site anaesthesia (General disorders) | 1 (2) | 0 (0)
Injection site bruising (General disorders) | 2 (13) | 4 (7)
Injection site discolouration (General disorders) | 5 (17) | 3 (12)
Injection site discomfort (General disorders) | 1 (38) | 2 (5)
Injection site erythema (General disorders) | 20 (112) | 22 (208)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 2 (4) | 1 (1)
Injection site induration (General disorders) | 7 (9) | 3 (17)
Injection site nodule (General disorders) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 7 (56) | 11 (102)
Injection site pruritus (General disorders) | 10 (36) | 11 (118)
Injection site swelling (General disorders) | 2 (8) | 5 (32)
Injection site warmth (General disorders) | 1 (44) | 3 (77)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04676724/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04676724/SAP_001.pdf